CLINICAL TRIAL: NCT02225639
Title: A Randomized, Double-blind Study of the Time Course of Response of PRC-063 in Adults With ADHD in a Simulated Adult Workplace Environment
Brief Title: PRC-063 in an ADULT Workplace Environment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rhodes Pharmaceuticals, L.P. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 063-008
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: ADHD; Adult
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRC-063 (Active Comparator)
  Interventions: Drug: PRC-063 25 mg; Drug: Placebo; Drug: PRC-063 35 mg; Drug: PRC-063 45 mg; Drug: PRC-063 55 mg; Drug: PRC-063 70 mg; Drug: PRC-063 85 mg; Drug: PRC-063 100 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: PRC-063 25 mg; Drug: Placebo; Drug: PRC-063 35 mg; Drug: PRC-063 45 mg; Drug: PRC-063 55 mg; Drug: PRC-063 70 mg; Drug: PRC-063 85 mg; Drug: PRC-063 100 mg

INTERVENTIONS:
Drug: PRC-063 25 mg — Oral 25 mg capsule - active
  Other Names: 25 mg capsule
Drug: Placebo — Oral placebo capsule
  Other Names: Placebo capsule
Drug: PRC-063 35 mg — Oral 35 mg capsule - active
  Other Names: 35 mg capsule
Drug: PRC-063 45 mg — Oral 45 mg capsule - active
  Other Names: 45 mg capsule
Drug: PRC-063 55 mg — Oral 55 mg capsule - active
  Other Names: 55 mg capsule
Drug: PRC-063 70 mg — Oral 70 mg capsule - active
  Other Names: 70 mg capsule
Drug: PRC-063 85 mg — Oral 85 mg capsule - active
  Other Names: 85 mg capsule
Drug: PRC-063 100 mg — Oral 100 mg capsule - active
  Other Names: 100 mg capsule

SUMMARY:
The primary objective of this study is to assess the time of onset and time course of efficacy over 16 hours of PRC-063 compared to placebo in adults diagnosed with ADHD in a simulated adult workplace environment (AWE) setting, as measured by the PERMP (an individually-adjusted math test) at pre-dose, 1.0, 2.0, 5.0, 8.0, 11.0, 14.0 and 16.0 hours post-dose.

DETAILED DESCRIPTION:
This is a randomized, double-blind, crossover, placebo-controlled, optimized-dose, phase 3 study to evaluate the safety and efficacy of PRC-063 (methylphenidate hydrochloride controlled-release capsules 25, 35, 45, 55, 70, 85 or 100 mg/day) in the treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) in adult subjects greater than or equal to 18 years of age and less than or equal to 60 years of age. After giving written informed consent, subjects will be screened to ascertain their suitability for the study according to the inclusion and exclusion criteria. The study will have four phases: (1) Screening and subsequent washout, if needed; (2) baseline and open-label dose optimization during which subjects will be titrated from a starting dose of 25 mg up to his/her final dose (25, 35, 45, 55, 70, 85 or 100 mg/day); (3) AWE sessions 1 and 2 in the adult analog setting following a practice session; and (4) 14-day safety follow-up. Subjects will be required to visit the clinic up to 10 times over a 9-week period.

ELIGIBILITY:
Inclusion Criteria:

* Must be male or non-pregnant female at least 18 years of age and less than or equal to 60 years of age.
* Must have an ADHD diagnosis, in attentive, hyperactive/impulsive or combined, as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) based on clinician assessment using multiple informants and a structured interview.
* Clinician-completed ADHD-5-RS total score must be equal to or greater than 24, as assessed at Visit 2a.
* Must be unsatisfied with his or her current pharmacological therapy for treatment of ADHD or not currently receiving pharmacological therapy for ADHD. Inclusion of subjects naïve to pharmacological therapy for ADHD is permitted.
* Female subjects must be one of the following: a. surgically sterile prior to screening; b. if of childbearing potential, abstinent or willing to use a reliable method of contraception, such as oral contraceptive, two barrier methods, a barrier method plus a spermicidal agent.
* Female subjects of Child-Bearing Potential (FOCP) must be a negative serum β-hCG pregnancy test at screening.
* Must have a minimum level of intellectual functioning, as determined by an Intelligence Quotient (IQ) score of 80 or above based on the KBIT-2.
* Mentally and physically competent to sign an informed assent document, in the case of the subject, and an informed consent document, in the case of the parent/guardian, indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Able and willing to comply with the study procedures for the entire length of the study, including a successful swallow test of an empty 100 mg capsule.

Exclusion Criteria:

* Having an allergy to methylphenidate or amphetamines or a history of serious adverse reactions to methylphenidate.
* Known to be non-responsive to methylphenidate treatment. Non-response is defined as methylphenidate use at various doses for a phase of at least four weeks at each dose with little or no clinical benefit in the last 10 years.
* Being diagnosed with or having a history of strokes, epilepsy, migraine headaches (greater than 1 instance every two months), glaucoma, thyrotoxicosis, tachyarrhythmias or severe angina pectoris or have serious or unstable medical illness. Subjects with controlled or stable asthma or diabetes will be permitted.
* Elevated blood pressure, defined as any values above 89 diastolic or 139 systolic, as assessed at Visit 1.
* Clinically significant ECG abnormalities, as assessed at Visit 1.
* Clinically significant laboratory abnormalities, as assessed at Visit 1.
* Currently receiving guanethidine, pressor agents, MAO inhibitors, coumarin anticoagulants, anticonvulsants (e.g., phenobarbital, phenytoin, primidone), phenylbutazone, tricyclic antidepressants (e.g., imipramine, desipramine), selective serotonin reuptake inhibitors (SSRIs) or herbal remedies (unless on a stable dose for 4 weeks).
* Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary heart disease, transient ischemic attack or stroke or other serious cardiac problems that may place the subject at increased vulnerability to the sympathomimetic effects of a stimulant drug.
* Subject has a known family history of sudden cardiac death or ventricular arrhythmia.
* Subjects who are currently considered a suicide risk by the investigator.
* Having a primary diagnosis of schizophrenia, schizoaffective disorder, primary affective disorder, schizotypal personality, major depression, bipolar disorder, generalized anxiety, borderline personality disorder, antisocial personality or another unstable psychiatric condition requiring treatment, as assessed by the structured interview conducted at Visit 1.
* Having a history or suspected physiological dependence within the past 5 years (excluding nicotine) on narcotic analgesics or other psychoactive drugs (including barbiturates, opiates, cocaine, cannabinoids, amphetamines and benzodiazepines).
* Excessive consumption of alcohol (consumes alcohol in quantities greater than 15 drinks per week; 1 drink is defined as 360 mL/12 oz. of beer, 120 mL/4 oz. of wine, or 30 mL/1 oz. of hard liquor), or history (within previous 6 months) of alcohol abuse.
* Currently (or within 30 days before the planned start of treatment) receiving an investigational drug or using an experimental medical device.
* Homeless.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Permanent Product Measure of Performance (PERMP) | Pre-dose, 1.0, 2.0, 5.0, 8.0, 11.0, 14.0 and 16.0 hours post-dose

SECONDARY OUTCOMES:
Observer-rated SKAMP | Pre-dose, 1.0, 2.0, 5.0, 8.0, 11.0, 14.0 and 16.0 hours post-dose
Clinician-administered ADHD-5-Rating Scale | 12.0 hours post-dose
Clinical Global Impressions of Improvement (CGI-I) | Pre-dose, 1.0, 2.0, 5.0, 8.0, 11.0, 14.0 and 16.0 hours post-dose
Subject-rated Conners' Adult ADHD Rating Scale (CAARS) | 12.0 hours post-dose
Self-report of the Pittsburgh Sleep Quality Index (PSQI) | Pre-dose, 1.0, 2.0, 5.0, 8.0, 11.0, 14.0 and 16.0 hours post-dose
Patient Satisfaction Survey (PSS) | Pre-dose, 1.0, 2.0, 5.0, 8.0, 11.0, 14.0 and 16.0 hours post-dose

OTHER OUTCOMES:
Occurrence of treatment-emergent adverse events and specific evaluation of blood pressure, heart rate, electrocardiogram (ECG), laboratory findings and physical examination (PE). | Controlled phase and 14-day safety followup
  AWE sessions 1 and 2 in the adult analog setting following a practice session; and (4) 14-day safety follow-up. Subjects will be required to visit the clinic up to 10 times over a 9-week period.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - AVIDA, Inc., Newport Beach, California
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada